CLINICAL TRIAL: NCT03718780
Title: Assessment of Continuous Measurement of Transcutaneous CO2 for Evaluation of Alveolar Dead Space During Exercise.
Acronym: TEASE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Metropole Savoie (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHMS18004
Record Dates: First submitted 2018-10-04; First posted 2018-10-24 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial; Chronic Heart Failure; Pulmonary Arterial Hypertension; Hyperventilation Syndrome; Healthy
Keywords: transcutaneous PtCO2; dead space; exercise test
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial; Pulmonary Arterial Hypertension | interventions — Blood Gas Monitoring, Transcutaneous; Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- A1: Patient in intensive care (Experimental): Patient in intensive care (n=10):
  in patients in the intensive care unit of the Centre Hospitalier Metropole Savoie (Chambéry, France), where repeated arterial blood gas analysis is routinely performed (Patients equipped for their usual care with an arterial catheter, enabling repeated arterial blood gas determination ).
  PaCO2 and Pt CO2 will be measured simultaneously at rest, and during conditions inducing PaCO2 modifications (ventilator settings modifications, or exercise as per routine rehabilitation) Comparison will be done between arterial PaCO2 and PtCO2
  Interventions: Other: simultaneous determination of PaCO2 and PtCO2
- A2: Healthy subjects (Experimental): Healthy subjects performing a voluntary hyperventilation, in the laboratory room where routine exercise testing is usually done.
  Comparison will be done between arterialized PaCO2 and PtCO2, at rest, and during an induced voluntary hyperventilation.
  Interventions: Other: Hyperventilation test; Other: Exercise test
- B1: Healthy subject (Experimental): Subjects, referred for exercise diagnostic testing, and whose results indicate normal cardiac and pulmonary exercise physiology.
  Measurement, throughout these exercise tests, of the alveolar dead space, and its kinetics, up to peak VO2, then during recovery, in the different conditions listed above. Alveolar dead space will be calculated using the continuous Pt CO2 values observed, and also with some intermittent PaCO2 measurement, done as per routine modus operandi (arterialized earlobe capillary drawn at rest, at ventilatory threshold, and at peak exercise). The values measured through PtCO2 and PaCO2 will be compared at these 3 time points.
  Interventions: Other: Exercise test
- B2: Chronic Obstructive Pulmonary Disease (Experimental): Measurement, throughout these exercise tests, of the alveolar dead space, and its kinetics, up to peak VO2, then during recovery, in the different conditions listed above. Alveolar dead space will be calculated using the continuous Pt CO2 values observed, and also with some intermittent PaCO2 measurement, done as per routine modus operandi (arterialized earlobe capillary drawn at rest, at ventilatory threshold, and at peak exercise). The values measured through PtCO2 and PaCO2 will be compared at these 3 time points.
  Interventions: Other: Exercise test
- B3: Interstitial Lung Disease (ILD) (Experimental): Measurement, throughout these exercise tests, of the alveolar dead space, and its kinetics, up to peak VO2, then during recovery, in the different conditions listed above. Alveolar dead space will be calculated using the continuous Pt CO2 values observed, and also with some intermittent PaCO2 measurement, done as per routine modus operandi (arterialized earlobe capillary drawn at rest, at ventilatory threshold, and at peak exercise). The values measured through PtCO2 and PaCO2 will be compared at these 3 time points.
  Interventions: Other: Exercise test
- B4: Chronic heart failure (CHF) (Experimental): Measurement, throughout these exercise tests, of the alveolar dead space, and its kinetics, up to peak VO2, then during recovery, in the different conditions listed above. Alveolar dead space will be calculated using the continuous Pt CO2 values observed, and also with some intermittent PaCO2 measurement, done as per routine modus operandi (arterialized earlobe capillary drawn at rest, at ventilatory threshold, and at peak exercise). The values measured through PtCO2 and PaCO2 will be compared at these 3 time points.
  Interventions: Other: Exercise test
- B5: Pulmonary Arterial Hypertension (PAH) (Experimental): Measurement, throughout these exercise tests, of the alveolar dead space, and its kinetics, up to peak VO2, then during recovery, in the different conditions listed above. Alveolar dead space will be calculated using the continuous Pt CO2 values observed, and also with some intermittent PaCO2 measurement, done as per routine modus operandi (arterialized earlobe capillary drawn at rest, at ventilatory threshold, and at peak exercise). The values measured through PtCO2 and PaCO2 will be compared at these 3 time points.
  Interventions: Other: Exercise test
- B6: inappropriate hyperventilation syndrome (Experimental): Measurement, throughout these exercise tests, of the alveolar dead space, and its kinetics, up to peak VO2, then during recovery, in the different conditions listed above. Alveolar dead space will be calculated using the continuous Pt CO2 values observed, and also with some intermittent PaCO2 measurement, done as per routine modus operandi (arterialized earlobe capillary drawn at rest, at ventilatory threshold, and at peak exercise). The values measured through PtCO2 and PaCO2 will be compared at these 3 time points.
  Interventions: Other: Exercise test

INTERVENTIONS:
Other: simultaneous determination of PaCO2 and PtCO2 — Patients in intensive care, equipped, for their routine clinical management, with an arterial catheter blood line, will have a simultaneous determination of PaCO2 and PtCO2:
  * 1) at rest; 2 arterial CO2/PtCO2 determinations will be carried out, 10 minutes apart
  * 2) During the muscular exercise part of their routine rehabilitation program (whatever it might be, limbs active mobilization, walking, etc...) : several arterial /PtCO2 samples will be collected during the first minutes of their muscular routine: 30 sec, 1 minute, 1 ½ minute, 2, 2 ½ , 3, 4, 5 minutes, 10 minutes (end of exercise). This will generate several couples of blood/transcutaneous CO2 determinations
  Arms: A1: Patient in intensive care
Other: Hyperventilation test — Repeated pairs of PtCO2 and PaCO2 (through arterialized capillary sampling), will be measured at the following timing: rest (0), then 30 sec post beginning of hyperventilation (breathing with accelerated frequency e.g. 30/min), 1 minute, 1 ½ minute 2, 2 ½ , 3, , 4, 5 minutes; recovery of this hyperventilation will be followed, for 5 minutes, with the PtCO2, during 3 minutes
  Arms: A2: Healthy subjects
Other: Exercise test — an exercise test, according to the routine protocol used in the clinic: initial phase of 3 minutes gentle pedaling (10 to 50 watts, according to subject capabilities), then stepwise increase in the workload, by increments of 20-40 watts every minute, until maximum tolerated workload (VO2max). Repeated pairs of PtCO2 and PaCO2 (through arterialized capillary sampling), will be measured at the following timing: rest -10 minutes, 0, then 30 sec post beginning of exercise, 1 minute, 1 ½ minute 2, 2 ½, 3 minutes, then 3 ½ minutes, then at mid-point of every step increase in workload, until maximum tolerated workload. Recovery will be followed with the PtCO2, for 5 minutes
  Arms: A2: Healthy subjects; B1: Healthy subject; B2: Chronic Obstructive Pulmonary Disease; B3: Interstitial Lung Disease (ILD); B4: Chronic heart failure (CHF); B5: Pulmonary Arterial Hypertension (PAH); B6: inappropriate hyperventilation syndrome

SUMMARY:
The study aim is to monitor, during exercise tests carried out in various conditions, the alveolar dead space, by means of continuous transcutaneous measurement of Pt CO2, which would be used as a surrogate for arterial PaCO2. Validity of this measurement needs to be assessed against arterial sampling (either arterial, or arterialized capillary), especially with regards to the lag time required by the CO2 diffusion from the arterial compartment (PaCO2) to the cutaneous one (PtCO2), in particular when rapid changes of CO2 might be induced by exercise.

The evaluation will be done in 2 different settings:

* intensive care patients, equipped, for their routine clinical care, with an arterial line; this allows for a precise timed comparison between PaCO2 and PtCO2 readouts;
* routine exercise test, where blood gas evaluation is done essentially by means of arterialized earlobe capillary sampling.

Following assessment of validity of the measurement (and the lag time PaCO2-PtCO2 which might be necessary to introduce as a correction), evolution of dead space during excise test will be tested in different conditions: Healthy subjects, patients with Chronic Obstructive Pulmonary Disease (COPD), chronic heart failure (CHF), hyperventilation, Pulmonary artery hypertension (PAH), or interstitial lung disease (ILD)

ELIGIBILITY:
Inclusion Criteria:

* Written and informed consent, and assent where required.
* Either:

Patients in intensive care, conscious and in stable hemodynamic condition, who are already equipped with an arterial line for blood gas analysis (as required by the routine practice in intensive care; no arterial line shall be inserted for the purpose of this study) (Part A1)

Or patients/subjects scheduled for routine cardio-pulmonary exercise testing. Among these, the following patients will be included: COPD, PAH, healthy subjects, hyperventilation, chronic cardiac failure, interstitial lung diseases (ILD) (Part A2 and Part B)

Exclusion Criteria:

* Non-French speaking patients/subjects
* Unstable hemodynamics
* Local cutaneous lesion or infection
* Arterial disease such as fistula
* Women with the following condition: pregnancy, breast feeding
* Persons deprived of liberty (according to article L1121-5 to L1121-8 of the French Public Health Code)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2019-02-22 (Actual); Primary Completion 2024-02-22 (Estimated); Study Completion 2024-02-22 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of Pt CO2 (transcutaneous CO2 partial pressure) measurement together with PaCO2 (arterial partial CO2 pressure) | at rest and during exercise/hyperventilation: 30 secondes, 1 minute, 1 ½ minute 2, 2 ½ , 3 , 4, 5 and 10 minutes.
  Part A: serial simultaneous measurements of Pt CO2 (transcutaneous CO2 partial pressure), and PaCO2 (arterial partial CO2 pressure), done
  1. during exercise
  2. during voluntary hyperventilation
Change from baseline by means of continuous measurement of alveolar dead space (VD/VT=(PaCO2-PECO2) /PaCO2), expressed as a percentage from 0% to 100 %) , during exercise test, in different clinical settings | continuous measurement: from rest throughout exercise test ( beginning of test, to maximum load (5-10 minutes), then throughout 5 minutes recovery.
  Part B: change from baseline with continuous alveolar dead space ( (VD/VT=(PaCO2-PECO2) /PaCO2), expressed as percentage from 0 to 100%) variation measurement, during exercise and recovery, in:
  * healthy subject
  * different patient categories: COPD at different stages, pulmonary artery hypertension, hyperventilation syndrome, cardiac failure, Interstitial Lung Disease). Establish patterns seen in these different conditions.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Service de pneumologie, Béthune
  - Service de pneumologie CHMS, Chambéry
  - Service de réanimation médicale - CHMS, Chambéry
  - Service de Pneumologie CHU Grenoble, La Tronche

IPD SHARING:
Plan to Share IPD: No